CLINICAL TRIAL: NCT00535223
Title: Group Based Exposure Therapy for Combat PTSD: RCT and Feasibility Study
Brief Title: Group Based Exposure Therapy for Combat-Related PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-010-06F
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Cognitive Behavior Therapy; Group therapy; Posttraumatic Stress Disorder; Randomized Controlled Trial; Treatment outcome; Veterans; War
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Based Exposure Therapy (Experimental): Behavioral:
  GBET is a 16-week program during which patients attend group therapy twice a week for three hours of group per day and are required to make two war trauma presentations to their group. These are recorded and the patients are required to listen to these recordings a minimum of 10 times. There are generally 10 patients per group and through the combination of making their own presentations, listening to recordings of these presentations, and hearing the presentations of the other nine group members, there are over 60 hours of exposure. Patients also learn about PTSD symptoms, sleep hygiene, specific stress/anger management techniques, and ways to cognitively restructure trauma-related thinking.
  Interventions: Behavioral: Group Based Exposure Therapy
- Present Centered Group Therapy (Experimental): Present Centered Group Therapy includes psych-education about PTSD and a problem solving "here and now" focus. This lasted for 16 weeks.
  Interventions: Behavioral: Present Centered Group Therapy

INTERVENTIONS:
Behavioral: Group Based Exposure Therapy — GBET is a 16-week program during which patients attend group therapy twice a week for three hours of group per day and are required to make two war trauma presentations to their group. These are recorded and the patients are required to listen to these recordings a minimum of 10 times. There are generally 10 patients per group and through the combination of making their own presentations, listening to recordings of these presentations, and hearing the presentations of the other nine group members, there are over 60 hours of exposure. Patients also learn about PTSD symptoms, sleep hygiene, specific stress/anger management techniques, and ways to cognitively restructure trauma-related thinking.
  Arms: Group Based Exposure Therapy
Behavioral: Present Centered Group Therapy — Present Centered Group Therapy includes psych-education about PTSD and a problem solving "here and now" focus.
  Arms: Present Centered Group Therapy

SUMMARY:
The purpose of this randomized controlled trial is to determine if Group Based Exposure Therapy (GBET) is more effective than treatment as usual in reducing the symptoms of war-related Posttraumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
Over 250,000 veterans with war-related PTSD were treated in the VA system in the VA system last year. Although the VA set up over 140 specialized PTSD programs and 206 Vet Centers to treat these veterans, a survey of practice patterns suggests that most VA PTSD treatment is not consistent with published treatment guidelines. This is mainly due to the very rare use of exposure therapy which is surprising considering that there is more empirical support for exposure therapy than for any other PTSD treatment. The failure to utilize evidence-based treatment may explain why studies have generally failed to support the efficacy of VA PTSD treatment. Group Based Exposure Therapy (GBET) is consistent with PTSD treatment guidelines and includes a large amount of exposure therapy. An open trial of 102 war veterans suggests that GBET produces clinically significant and lasting PTSD symptom reductions, as measured by the Clinician Administered PTSD Scale (CAPS), with a large effect size of 1.20 (generalized d). Clinically significant symptoms reductions, defined as a reduction in total CAPS score of 10 or more points, were found in 81 percent of patients. These symptom reductions were maintained on 6-month post-treatment assessments for most patients. Self-report measures of depression, anger, suicidal ideation and PTSD were also significantly reduced when pre-treatment measures were compared to post-treatment scores. This magnitude of symptom change has rarely been reported with VA war-related PTSD patients and there was a low dropout rate (>3%). Caution should be used in interpreting these unusual findings due to the treating clinicians conducting study assessments. Unconscious bias or a desire by patients to please their therapists may have affected outcomes. GBET is a 16-week program during which patients attend group therapy twice a week for three hours of group per day and are required to make two war trauma presentations to their group. These are recorded and the patients are required to listen to these recordings a minimum of 10 times. There are generally 10 patients per group and through the combination of making their own presentations, listening to recordings of these presentations, and hearing the presentations of the other nine group members, there are over 60 hours of exposure. Patients learn about PTSD symptoms, sleep hygiene, specific stress/anger management techniques, and ways to cognitively restructure trauma-related thinking. Although these findings are encouraging critical questions remain about the generalizability of GBET. The three primary questions are: 1) would similar outcomes be found with the more rigorous test of a randomized controlled trial, 2) can new psychotherapists produce similar outcomes, and 3) can similar outcomes be found at other sites. The proposed study would take the next step by conducting the first controlled trial in which 88 veterans with war-related PTSD will be randomly assigned to either GBET or Treatment as Usual control condition (44 per condition). GBET treatment would be provided by four psychotherapists without prior GBET experience. Independent Assessors blind to treatment condition would assess patients prior to treatment, at post-treatment, 6-months post-treatment and one year post-treatment using CAPS and other standardized measures. If GBET is supported, multi-site study will be proposed to investigate the third primary question.

Potential Impact on Veteran Health Care: GBET was developed within a specialized PTSD program, by VA clinicians working with war veterans and has been a primary mode of treatment within this program for over three years. Most VA PTSD programs have staffing similar to the one the developed GBET and many have more staff. GBET is manualized and could be adopted easily by other VA PTSD programs and Vet Centers. The proposed study would serve as a feasibility study for a multi-site study. If a multi-site study found that GBET produced superior treatment outcomes to those currently in use, it could have a direct impact on the lives of a large number of veterans by leading to better PTSD treatment within the VA.

ELIGIBILITY:
Inclusion Criteria:

1. Male veterans diagnosed with war-related PTSD as assessed by the CAPS. Patients must provide a DD214 or other documentation of war exposure.
2. Patients must have the ability to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments (as evident by the ability to pass informed consent test, to fill out self-report assessment measures and to respond appropriately during the clinical interview).
3. Patients must be either stable on psychotropic medication (defined as no additional psychotropic medications or significant increases in previously prescribed psychotropic medications for a period of at least three months) or not on psychotropic medication.
4. Patients must be currently in treatment within the Mental Health Clinic (MHC) of the Atlanta VA Medical Center for a minimum of four months prior to participation. This would insure adequate psychiatric coverage and case management. If a change in medication were needed during the study, it would be made. Such changes would be tracked for analysis if they occur in a significant number of patients.
5. Patients must have the support of their current Mental Health Clinic Treatment Team to participate in the study.

Exclusion Criteria:

Exclusion criteria are intended to exclude patients who might be harmed by study participation and to yield as ecologically valid a sample as possible.

1. Patients with current or history of mania or schizophrenia would be excluded because the stress of exposure therapy may precipitate an increase in symptoms of these co-morbid conditions that could interfere with the patient's ability to benefit from treatment.
2. Patients suffering from current active psychosis, active mania, or sufficient mental impairment, as assessed by a Mini Mental State Exam score below 24, which would prevent the patient from providing valid consent or participating safely or understanding the treatment.
3. Patients with current, prominent suicidal ideation. All patients would be screened for suicidal ideation and intention by the RC in the initial screening and again by the IA in the initial assessment through a brief clinical interview. A BDI #9 score above 3 would prompt a more in-depth inquiry concerning suicidal thoughts and intentions during the initial assessment.
4. Patients who currently meet diagnostic criteria for substance abuse or dependence or have met such criteria during the previous three months (as measured by the clinical interview and the Kreek-McHugh-Schluger-Kellogg scale (50)).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-07; Primary Completion 2010-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ready, PhD MS, Principal Investigator — VA Medical Center, Decatur
Locations (1):
- VA Medical Center, Decatur, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 male, Vietnam era veterans referred for PTSD treatment were informed about the study, 98 consented to participate, 11 dropped out before randomized, 6 were excluded due to (3)psychosis or manic symptoms and 3 did not have PTSD. 40 were assigned to PSGT and 41 to GBET. One assigned to GBET, dropped out during the first week and was replaced.
Pre-assignment Details: Participants had been referred to an outpatient PTSD program, were first screened by the staff of that program and if judged to be appropriate for intensive PTSD treatment were informed about the study. They could request to be screened for the study or go directly into one of the treatments provided by the PTSD program.
Period: Overall Study
Arm/Group | Group Based Exposure Therapy | Present Centered Group Therapy
Started | 41 (Patients were randomized in cohorts of ten.) | 40 (Patients were randomized in cohorts of ten.)
Completed | 37 | 39
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Based Exposure Therapy | Present Centered Group Therapy | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 37 | 77
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 61.41 [55 to 68] | 61.38 [55 to 69] | 61.40 [55 to 69]
Sex/Gender, Customized [Number; unit: participants]
  Male | 41 | 40 | 81
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: This is an interview regarding the frequency and intensity of each of the 17 PTSD symptoms found in DSM IV and includes information about the degree to which these symptoms are interfering with functioning. This interview includes that clinician rating the participants responses for both the frequency of each symptom and the intensity of each symptom on a scale of zero to four. A score of 0, best possible score, would indicate that the participant is no longer reporting any of the 17 DSM IV symptoms of PTSD. The worse possible score is 136, this would indicate that a participant was reporting every symptoms of PTSD occurring daily or almost daily and that each symptom is causing the most extreme level of distress.
Time Frame: Pre treatment, Post treatment (16 weeks) and One year post treatment
Population: Pre-tx Post-tx 1-yr F.U. N M SD Range N M SD Range N M SD Range GBET 41 82.44 15.09 55-107 41 71.73 20.55 34-105 35 69.29 20.71 24-107 PCGT 40 81.18 14.31 52-109 40 75.43 23.01 18-122 33 71.03 22.80 37-121
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group Based Exposure Therapy: See below
  Group Based Exposure Therapy: GBET is a 16-week program during which patients attend group therapy twice a week for three hours of group per day and are required to make two war trauma presentations to their group. These are recorded and the patients are required to listen to these recordings a minimum of 10 times. There are generally 10 patients per group and through the combination of making their own presentations, listening to recordings of these presentations, and hearing the presentations of the other nine group members, there are over 60 hours of exposure. Patients also learn about PTSD symptoms, sleep hygiene, specific stress/anger management techniques, and ways to cognitively restructure trauma-related thinking.
- Present Centered Group Therapy: The group met twice a week for 16 weeks for 90 minutes per session. The focus was on dealing with problem solving in the here and now while avoiding traumatic material.
Arm/Group | Group Based Exposure Therapy | Present Centered Group Therapy
Number analyzed (Participants) | 41 | 40
units on a scale
  Pre treatment | 82.4 (15.09) | 81.18 (14.31)
  Post treatment[ | 71.73 (20.55) | 75.43 (23.01)
  one yr post tx (N= 35 GBET & N=33 PCGT | 69.29 (20.71) | 71.03 (22.80)

2. Secondary Outcome: Posttraumatic Cognitions Inventory (PTCI)
Description: This 36 item self-report measure is designed to assess the degree to which a participant agrees with thoughts and beliefs that have been found to be common for individuals who suffer from PTSD. Each item is rated between 1 ( Totally Disagree) to 7 ( Totally Agree). The best score would be 36, indicating that the participant totally did not agree with any of the thoughts that have been associated with PTSD. The worse score would be 252, which would indicate that the participant totally agreed with all of the cognitions that have been associated with PTSD
Time Frame: Pre-treatment, Post-Treatment (16 weeks) and One year Post Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Based Exposure Therapy | Present Centered Group Therapy
Number analyzed (Participants) | 41 | 40
units on a scale
  Pre treatment | 145.45 (30.19) | 135.29 (35.22)
  Post treatment | 130.07 (34.84) | 139.58 (40.52)
  One yr post tx (N=35 GBET & N= 33 PCGT | 127.36 (40.48) | 140.57 (34.45)

ADVERSE EVENTS:
Time Frame: For the whole four years of the study.
Groups:
- Group Based Exposure Therapy: Group Based Exposure Therapy. No serious adverse events occurred in response to this treatment.
- Present Centered Group Therapy: Present Centered Group Therapy. No serious adverse events occurred in response to this treatment.
Arm/Group | Group Based Exposure Therapy | Present Centered Group Therapy
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No